CLINICAL TRIAL: NCT02619552
Title: Impact of Medical Treatment on Sexual Function in Patients With Crohn's Disease
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Vanderbilt University (Other); Milton S. Hershey Medical Center (Other); Mercy Medical Center (Other)
Responsible Party: Principal Investigator, Raymond Cross, Professor of Medicine, University of Maryland, Baltimore
Other Study IDs: HP-00050472
Record Dates: First submitted 2015-10-28; First posted 2015-12-02 (Estimated); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Crohn's Disease; IBD
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab; Adalimumab; Certolizumab Pegol; Steroids; Prednisone; Budesonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Anti-TNF (Remicade, Humira or Cimzia) for luminal CD: All participants are required to undergo study visits at baseline, 2 months, and 6 months in addition to any other routine visits. Sexual function, body image, disease activity, quality of life, and depression scores will be measured at baseline and at each study visit during the 6-month study.
  Interventions: Drug: Anti-TNF
- Anti-TNF (Remicade, Humira or Cimzia)for perianal CD: All participants are required to undergo study visits at baseline, 2 months, and 6 months in addition to any other routine visits. Sexual function, body image, disease activity, quality of life, and depression scores will be measured at baseline and at each study visit during the 6-month study.
  Interventions: Drug: Anti-TNF
- Steroid (Prednisone or budesonide) for luminal CD: All participants are required to undergo study visits at baseline, 2 months, and 6 months in addition to any other routine visits. Sexual function, body image, disease activity, quality of life, and depression scores will be measured at baseline and at each study visit during the 6-month study.
  Interventions: Drug: Steroids

INTERVENTIONS:
Drug: Anti-TNF — All participants in this arm receive an anti-TNF for the treatment of luminal CD. They are required to undergo study visits at baseline, 2 months, and 6 months in addition to any other routine visits. Sexual function, body image, disease activity, quality of life, and depression scores will be measured at baseline and at each study visit during the 6-month study.
  Other Names: Remicade, Humira, Cimzia
  Groups: Anti-TNF (Remicade, Humira or Cimzia) for luminal CD
Drug: Anti-TNF — All participants in this arm receive an anti-TNF for the treatment of perianal CD. They are required to undergo study visits at baseline, 2 months, and 6 months in addition to any other routine visits. Sexual function, body image, disease activity, quality of life, and depression scores will be measured at baseline and at each study visit during the 6-month study.
  Other Names: Remicade, Humira, Cimzia
  Groups: Anti-TNF (Remicade, Humira or Cimzia)for perianal CD
Drug: Steroids — All participants in this arm receive steroids for the treatment of luminal CD. They are required to undergo study visits at baseline, 2 months, and 6 months in addition to any other routine visits. Sexual function, body image, disease activity, quality of life, and depression scores will be measured at baseline and at each study visit during the 6-month study.
  Other Names: Prednisone, Budesonide
  Groups: Steroid (Prednisone or budesonide) for luminal CD

SUMMARY:
Crohn's disease is a chronic inflammatory condition of the intestines that causes abdominal pain, diarrhea, tunnels around the anus (fistulas), and extraintestinal symptoms. Effective medical treatments exist to treat the disease; however they can have significant side effects.

Previous studies have shown that sexual function is impaired in patients with Crohn's disease. It is likely that both the symptoms related to the disease, medications used to treat the disease, and surgery all impair sexual function in a variety of ways. For example, body image may be impaired, patients may be worried about bowel incontinence or unpleasant odors associated with diarrhea, patients may have significant pelvic pain secondary to perianal fistulas, or they may have painful intercourse from adjacent inflammation or scarring in the pelvis. The impact of medical treatment on patient's ability to regain sexual function is not known.

The investigators propose a 6 month study to compare sexual function before and after treatment in patients with Crohn's disease about to initiate therapy with an anti-TNF drug for treatment of perianal fistula or intestinal Crohn's or about to initiate therapy with steroids.

The investigators anticipate that the investigators will show that therapy with an anti TNF agent will result in a more rapid and greater return of sexual function than steroids. This information will be important to help counsel patients about the optimal treatment to begin for treatment of their Crohn's disease. Furthermore, it would be the first study to evaluate the impact of medical therapy on sexual function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease confirmed by standard criteria
* Active luminal Crohn's disease defined by an HBI score of >4 or with draining perianal Crohn's disease a) Active perianal Crohn's disease defined a presence of draining perianal fistula on physical exam19
* Patients with active luminal Crohn's disease must be initiating treatment with an anti-TNF agent (Remicade, Humira, Cimzia, or Simponi) or a steroid (prednisone, Entocort, or Uceris).
* Patients with active perianal disease must be initiating therapy with an anti-TNF agent (Remicade, Humira, Cimzia, or Simponi).
* Can understand written instructions in English

Exclusion Criteria:

* Previous primary non-response to an anti-TNF
* Uncontrolled medical or psychiatric disease (a. Degenerative neurologic condition, b.Unstable angina, c.Class III/IV congestive heart failure, d.Severe asthma or chronic obstructive pulmonary disease, e.Symptomatic peripheral vascular disease, f. Chronic renal insufficiency (creatinine > 2.0), g. Malignancy within the last 3 years (excluding squamous or basal cell cancers of the skin), h. Poorly controlled depression, mania, and schizophrenia, i. Active infection, j. Acquired immunodeficiency syndrome)
* Inability to adhere to the protocol
* Need for imminent surgery other than an exam under anesthesia
* Under 18 years of age.
* Pregnancy
* Use of concurrent prednisone >30 mg per day in the anti-TNF groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators are planning a study with 60 experimental participants and 30 control participants. The investigators will recruit participants from multiple referral centers for IBD with an existing population of nearly 5,000 patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Sexual Function | 6 months
  Sexual Function Questionnaire
Assessment of Disease Activity | 6 months
  Harvey Bradshaw Index
Assessment of Quality of Life | 6 months
  Short Inflammatory Bowel Disease Questionnaire
Assessment of Body Image | 6 months
  Body Image Scale
Assessment of Depression | 6 months
  PHQ 9
Assessment of Perianal Disease Activity | 6 months
  Perianal Disease Activity Index

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Cross, MD, MS, Principal Investigator — University of Maryland, Baltimore
Locations (4):
- United States (4):
  - Mercy Medical Center, Baltimore, Maryland
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee